CLINICAL TRIAL: NCT00440622
Title: A Multicenter Randomized Phase III Study of Gemcitabine Plus Herceptin Combination Versus the Capecitabine Plus Herceptin Combination in Pretreated Patients With HER-2 Positive Metastatic Breast Cancer
Brief Title: Study of Gemcitabine and Herceptin Versus Xeloda and Herceptin in HER-2 (+) Metastatic Breast Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/03.09
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: Cancer; Metastatic Breast cancer; Her-2 expression; Gemcitabine; Capecitabine; Herceptin
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Gemcitabine; Trastuzumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): GHer
  Interventions: Drug: Gemcitabine; Drug: Herceptin
- 2 (Experimental): CapHer
  Interventions: Drug: Herceptin; Drug: Capecitabine (Xeloda)

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine at the dose of 1250 mg/m2 IV on day 1 every 3 weeks for 6 cycles
  Other Names: Gemzar
  Arms: 1
Drug: Herceptin — Herceptin 8 mg/Kg (90 min IV) on day 1 for the first cycle and 6 mg/Kg for the 5 remaining cycles over a 30 min IV
Drug: Capecitabine (Xeloda) — Capecitabine at the dose of 1250 mg/m2 b.i.d p.o on day 1-14 every 3 weeks 6 cycles
  Other Names: Xeloda
  Arms: 2

SUMMARY:
The optimal treatment for pretreated patients with metastatic breast cancer has not been established. Gemcitabine and capecitabine are two active agents in this setting. For women with Her-2 positive breast cancer, combinations of either gemcitabine or capecitabine (Xeloda) plus Herceptin has been proved active and well tolerated.

DETAILED DESCRIPTION:
This trial compares the efficacy of the combinations gemcitabine plus Herceptin versus capecitabine (Xeloda) plus Herceptin in pretreated patients with metastatic HER-2 positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Histologically confirmed metastatic breast adenocarcinoma (stage IV) without any prior chemotherapy received
* HER-2 overexpression 2+ or 3+ using IHC or FISH +
* Measurable disease
* At least one prior chemotherapy regimen
* Not in a prior irradiation field
* No patients with brain metastatic disease who has not been irradiated or uncontrolled brain metastatic disease after irradiation
* No more than 25% of myeloproductive bone marrow irradiated. More than 4 weeks since prior radiotherapy and recovered
* Age 18 - 75 year old
* Performance status (WHO) 0-2
* Life expectancy more than 12 weeks
* Absolute neutrophil count > 1500/mm^3, platelet count > 100000/mm^3, hemoglobin > 9 gr/mm^3)
* Adequate liver (bilirubin < 2 mg/dL, SGOT/SGPT < 2 times upper limit of normal, ALP < 3 times upper limit of normal, creatinine < 1.5 upper limit of normal
* Adequate cardiac function (LVEF > 50%)

Exclusion Criteria:

* Pregnant or nursing
* Positive pregnancy test
* Concurrent agents ketoconazole, macrolide antibiotics, zidovudine which may induce P-450 cytochrome
* Motor or sensory neuropathy > grade 1 according to NCIC toxicity criteria
* History of allergic reaction attributed to docetaxel
* Psychiatric illness or social situation that would preclude study compliance
* Other concurrent uncontrolled illness
* Other invasive malignancy within the past 5 years except cured basal cell skin carcinoma and cervical carcinoma in situ

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2003-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) between the two treatment arms | 1 year

SECONDARY OUTCOMES:
Overall survival | 1 year
Toxicity profile | During the time of chemotherpy

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete
Locations (9):
- Greece (9):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki